CLINICAL TRIAL: NCT05511636
Title: A Randomized Controlled Trial To Compare The Outcome Of High Flow Oxygen Versus Conventional Oxygen In Extubated Patients After Lung Resection.
Brief Title: Comparing The Outcome Of High Flow Oxygen Versus Conventional Oxygen In Extubated Patients After Lung Resection.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cardiothoracic academy
Record Dates: First submitted 2022-07-05; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Resection; Oxygen Therapy
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- those that receive the conventional oxygen (Experimental): This study will be conducted on 180 patients who will be undergoing lung resection (wedge resection, segmentectomy, metastasectomy, lobectomy, or pneumonectomy) surgery at the Cardiothoracic department, Ain Shams University Hospitals; patients are to be extubated intraoperative, and at the ICU will be given HFNC . The endpoints of the study are to investigate whether high-flow nasal cannula oxygen therapy is superior to conventional oxygen therapy for reducing hypoxemia and postoperative pulmonary complications in extubated patients after lung resection.
  Interventions: Other: Oxygen therapy
- those that receive the high flow oxygen therapy. (Experimental): This study will be conducted on 180 patients who will be undergoing lung resection (wedge resection, segmentectomy, metastasectomy, lobectomy, or pneumonectomy) surgery at the Cardiothoracic department, Ain Shams University Hospitals; patients are to be extubated intraoperative, and at the ICU will be given standard oxygen therapy . The endpoints of the study are to investigate whether high-flow nasal cannula oxygen therapy is superior to conventional oxygen therapy for reducing hypoxemia and postoperative pulmonary complications in extubated patients after lung resection.
  Interventions: Other: Oxygen therapy

INTERVENTIONS:
Other: Oxygen therapy — This study will be conducted on 180 patients who will be undergoing lung resection (wedge resection, segmentectomy, metastasectomy, lobectomy, or pneumonectomy) surgery at the Cardiothoracic department, Ain Shams University Hospitals; patients are to be extubated intraoperative, and at the ICU we will be comparing HFNC to standard oxygen therapy. The endpoints of the study are to investigate whether high-flow nasal cannula oxygen therapy is superior to conventional oxygen therapy for reducing hypoxemia and postoperative pulmonary complications in extubated patients after lung resection.
  Other Names: oxygen

SUMMARY:
Conventional oxygen therapy (COT) is the main supportive treatment administered to patients postoperative after planned extubation and has conventionally been delivered using nasal prongs, cannula or masks. However, the maximal oxygen flow rates that these devices can deliver are limited. Being diluted by the ambient air which reduces the fraction of inspired oxygen is not only the main concern, but also COT is difficult to meet the requirements of heating and humidification in extubated patients. Yu Y, et al. (2017)

High-flow nasal cannula (HFNC) can supply a mixture of air and oxygen via a heated and humidified circuit at a very high flow. It can provide almost pure oxygen with a FiO2 of approximately 100% and a maximal flow rate up to 60 L/min. The use of a HFNC may generate a positive airway pressure, ameliorate oxygenation and dyspnea, reduce the respiratory rate and work of breathing, and improve comfort. Yu Y, et al. (2017)

Few studies were conducted in the past 5 years; and the effect of HFNC therapy compared to COT in patients after planned extubation remains inconclusive. This study will be done to compare the usage of HFNC as an alternative to the conventional oxygen therapy following extubation for patients undergoing pulmonary resection. Youfeng Zhu, et al. (2019)

DETAILED DESCRIPTION:
Postoperative interventions effective in the reduction of pulmonary complications include good pain control, incentive spirometry, oxygen therapy, intermittent continuous positive airway pressure (CPAP), and early mobilization. Simple techniques such as incentive spirometry and patient positioning have proven to be ineffective in countering atelectasis, which can occur postoperatively in as many as 90% of patients. Noninvasive ventilatory support in the form of CPAP has been used as both a prophylactic and therapeutic intervention to improve ventilation in postoperative patients. Although CPAP may prevent pulmonary complications, it is uncomfortable for patients because it is applied by a tight-fitting mask, and patients may complain of difficulty with communication, eating and drinking, and mobilization, and consequently compliance is often poor. Bilal M. Ansari, et al. (2016)

Conventional oxygen therapy via nasal prongs or a facemask can supplement oxygen administration, in some of the patients specially those who have lobectomy, it is ineffective in compensating for loss in lung volume or in maintaining gas exchange. High-flow nasal cannula oxygen (HFNC) mainly delivers a flow-dependent positive airway pressure and improves oxygenation by increasing end-expiratory lung volume. It is considered to have a number of physiological advantages compared with other standard oxygen therapies, including the provision of positive end-expiratory pressure (PEEP), constant FiO2, and good humidification. More importantly, it can reduce the anatomical dead space. Youfeng Zhu, et al. (2019)

HFNC can be widely employed for patients of all age groups in several types of respiratory failure from preterm infants to adults and is broadly used in ICU because of the ease of use, tolerability, and safety. Youfeng Zhu, et al. (2019) HFNC systems now are increasingly being utilized, as when compared to regular nasal cannula and facemask oxygen, HFNC appears to be linked to decreased level of respiratory complications and hypoxemia after lung resection. Yu Y, et al. (2017)

Few studies were conducted comparing different modalities of oxygen therapy; however, the answer of this question is still controversial. Is HFNC should be used as an alternative to the conventional oxygen therapy for patients undergoing lung resection following extubation ?

ELIGIBILITY:
Inclusion Criteria:

* • Patients undergoing elective lung resection, including lobectomy, wedge resection, segmentectomy, metastasectomy; open thoracotomy or video-assisted thoracoscopic surgery (VATS)

Exclusion Criteria:

* • Age below 10 years and above 80 years, as this age range was the age in the 2 pervious studies in literature.

  * Immunocompromised patients.
  * Pregnant females.
  * Patients with history of obstructive sleep apnea.
  * Tracheostomized patients.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
HFNC is superior to conventional oxygen for reducing hypoxemia [arterial partial pressure of oxygen/fraction of inspired oxygen] < 300) and postoperative pulmonary complications occurring within 30 days in extubated patients after lung resection. | 120 weeks
  patients were extubated intraoperative, and at the ICU we compared HFNC to standard oxygen therapy. Postoperative pulmonary function expressed as ppoFEV1 (predicted postoperative forced expiratory volume in one second) was prognosticated preoperatively using spirometry. Oxygen therapy was delivered for at least 48 hours, and if any patient needed more time on oxygen therapy; it was maintained and patients were allowed to be transferred from control group to study group if needed, but didn't happen.
  HFNC oxygen therapy group (HFNCG) received a flow rate of 35 to 60 L/min and FiO2 was titrated (from 45% to 100%) by the treating clinician to maintain a peripheral oxygen saturation (SpO2) of 95% or more. The conventional oxygen therapy group (COG) received oxygen via either nasal prongs or facemask with oxygen flow titrated by the bedside clinician to maintain a SpO2 of 92% or more.

CONTACTS AND LOCATIONS:
Overall Officials: ahmed t. hussain kamel, MSC, Principal Investigator — ainshams uU
Locations (1):
- Ainshams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Yes

REFERENCES:
- [Background] Yu Y, Qian X, Liu C, Zhu C. Effect of High-Flow Nasal Cannula versus Conventional Oxygen Therapy for Patients with Thoracoscopic Lobectomy after Extubation. Can Respir J. 2017;2017:7894631. doi: 10.1155/2017/7894631. Epub 2017 Feb 19. PMID 28298878